CLINICAL TRIAL: NCT04696224
Title: Comparative Use of Tranexamic Acid Intravenous and Topical Application in the Treatment of Intertrochanteric Fractures With Proximate Femoral Nail
Brief Title: Comparative Use of Tranexamic Acid Intravenous and Topical Application in Intertrochanteric Fractures With PFNA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Vale do Sapucai (Other)
Responsible Party: Principal Investigator, Carlos Delano Mundim Araujo, Professor, Universidade do Vale do Sapucai
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 38830520.3.0000.5102
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Hemorrhage; Fracture Femur
Keywords: Tranexamic acid; Hemorrhage; Hip fractures; blood transfusion
MeSH Terms: conditions — Hemorrhage; Femoral Fractures; Hip Fractures | interventions — Tranexamic Acid; Surgical Procedures, Operative; Saline Solution

STUDY DESIGN:
Intervention Model Description: Primary, analytical, prospective, interventional, double-blind, controlled, randomized study in humans.
Who Masked: Participant, Investigator
Masking Description: For randomization, the computer generated random sequence (BIOESTAT 5.0) will be used. The allocation concealment will be guaranteed by the consecutive opening of numbered, opaque sealed envelopes, after anesthetic induction, opened by the anesthetist, who will be responsible for the intravenous administration and for instructing the nurse of the room about what should be placed in a vat for topical use: saline or tranexamic acid. The orthopedic medical team and the patient will not be aware of which of these will be used intravenously or topically (double blind). The envelopes opened by the anesthetist will have a card written: "intravenous" or "local" or "placebo".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- INTRAVENOUS (Active Comparator): 30 patients who will receive 15mg / kg of TXA intravenous in 100ml salina solution (0,9%), after anesthetic induction and before incising the skin (administered in 10 minutes). For masking purposes, these patients will also receive at the end of the surgery, and before performing the plan closure, a compress soaked in 80ml of saline solution (0.9%), which will fill all the plans of the incision, and will be kept for 5 minutes.
  Interventions: Drug: Tranexamic acid
- LOCAL (Active Comparator): 30 patients who, at the end of the surgery, and before the suture in layers, will receive a compress soaked in a solution of 1.5 g of tranexamic acid (six ampoules of Transamin®, Zydus Nikkho) diluted in 50 ml of saline solution (0.9 %) (total volume of 80ml), which will fill all the plans of the incision and will be maintained for 5 minutes. For masking purposes, these patients will also receive 100ml of saline solution (0.9%) after anesthetic induction and before incising the skin.
  Interventions: Drug: Tranexamic acid
- PLACEBO (Placebo Comparator): 30 patients who will not receive the TXA, but will receive a 100ml intravenous saline solution 0,9% after anesthetic induction and before incising the skin (such as group 1) and a compress soaked in saline solution as used in group 2.
  Interventions: Other: Saline solution

INTERVENTIONS:
Drug: Tranexamic acid — The surgical technique consists in patient in supina position with previous reduction with lower limb traction (on a traction table or manual) associated or not with the use of percutaneous reduction clamps. Longitudinal lateral incision of 3-5 cm proximal to the greater trochanter, approximately 5 cm long, will be performed. After the skin and subcutaneous incision, the fascia lata will be incised in the same direction, with exposure of the gluteal muscles and the proximal femur. The awl will be introduced at the tip of the greater trochanter and then, at the same location, an intramedullary guidewire, towards the proximal shaft, crossing the fracture. A 3 cm incision to the thigh and inferior to the initial incision with template to introduce the screw in the center of the femoral head. Then, a 2cm incision will be made at the distal end of the nail, and a hole in the femur for the distal lock in dynamic nail hole with a 4.5mm drill where a cortical screw will be inserted.
  Other Names: surgery
  Arms: INTRAVENOUS; LOCAL
Other: Saline solution — 30 patients who will not receive the TXA, but will receive a 100ml intravenous saline solution 0,9% after anesthetic induction and before incising the skin (such as group 1) and a compress soaked in saline solution as used in group 2
  Arms: PLACEBO

SUMMARY:
An intertrochanteric (ITF) trochanteric fracture of the femur is an exclusively extra capsular fracture in which the fracture line extends from the greater trochanter to the lesser trochanter. Its incidence has increased significantly over the past decades and is expected to double in the next 25 years, with an important global economic impact . It affects women in the seventh and eighth decades of life, an age group older than femoral neck fractures. For this reason, the mortality of intertrochanteric fractures is twice that of the femoral neck.

The treatment is surgical, in which the objective is the stable internal fixation and the patient's early ambulation.

Functional outcomes and treatment mortality are related including factors perioperative anemia and blood loss.Even so, even with these precautions, blood loss in this surgical procedure appears to be greater than expected, with blood loss of the order of 2100ml.

Blood loss management and the inherent risks of anemia can be circumvented with blood transfusion. However, blood transfusion is not without risks and complications, such as hypersensitivity and hemolytic reactions, cardiac overload, infectious diseases. Homologous transfusions are associated with prolonged hospital stay, increased costs and increased patient morbidity and mortality.

So, alternatives have been used to avoid the use of blood such as saline solutions, use of erythropoietin and antifibrinolytic agents . Tranexamic acid (TXA) is a drug that interferes with fibrinolysis, in use for more than 50 years in surgery, particularly in cardiac surgery.

Only recently, TXA has sparked interest in orthopedic surgeries. Studies have shown the effectiveness and safety of TXA at FIT, but presented different forms of administration (intravenous, topical, infiltrative) . Despite promising results to contain bleeding in elective orthopedic surgery and fractures, in daily practice, TXA is not very popular, especially in fractures, and has not been used routinely by all doctors. Studies have not been found in the literature about the topical use of TXA compared to intravenous use in FIT.

DETAILED DESCRIPTION:
An intertrochanteric (ITF) trochanteric fracture of the femur is an exclusively extra capsular fracture in which the fracture line extends from the greater trochanter to the lesser trochanter. Usually, it is an isolated fracture, related to osteoporosis, which occurs due to low-energy trauma such as a fall during gait. It is the most common fracture of the proximal femur. Its incidence has increased significantly over the past decades and is expected to double in the next 25 years, with an important global economic impact . It affects women in the seventh and eighth decades of life, an age group older than femoral neck fractures. For this reason, the mortality of intertrochanteric fractures is twice that of the femoral neck.

The treatment is surgical, in which the objective is the stable internal fixation and the patient's early ambulation. The most used materials are plates with dynamic compression screws (Dinamic Hip Screw-DHS) and intramedullary nails (specifically cephalomedullary nails or Proximate femoral nail (PFN). Patients who have suffered this fracture are at high risk for cardiovascular, pulmonary, infections and thrombosis. About a third of patients die in the first year after the injury, approximately 50% become incapable of walking alone or climbing stairs and 20% need permanent home care.

Functional outcomes and treatment mortality are related including factors perioperative anemia and blood loss. In order to prevent blood loss, many strategies have been taken, such as closed or percutaneous fracture reduction and surgical approach with minimally invasive techniques such as fixation with short intramedullary nails (PFN). Even so, even with these precautions, blood loss in this surgical procedure appears to be greater than expected, with blood loss of the order of 2100ml. It was also observed that surgeons underestimate the amount of blood lost in the perioperative period, having estimated a median difference of 1473ml between the apparent blood loss and the one that actually occurred with the use of cephalomedullary nails. Blood loss in ITF is greater than in femoral neck fractures and more often requires blood transfusions.

Blood loss management and the inherent risks of anemia can be circumvented with blood transfusion. However, blood transfusion is not without risks and complications, such as hypersensitivity and hemolytic reactions, cardiac overload, infectious diseases. Homologous transfusions are associated with prolonged hospital stay, increased costs and increased patient morbidity and mortality. Some surgeries may need to wait for the blood supply to be replenished and patients in need of phenotyped blood find it even more difficult and may wait days to weeks before finding their proper blood type.

So, alternatives have been used to avoid the use of blood such as saline solutions, use of erythropoietin and antifibrinolytic agents . Tranexamic acid (TXA) is a drug that interferes with fibrinolysis, in use for more than 50 years in surgery, particularly in cardiac surgery.

Only recently, TXA has sparked interest in orthopedic surgeries. Then it has been used in spine surgery, and joint replacement, without reports of complications. Despite extensive studies on its use in elective orthopedic surgeries, and its high safety profile, there are few studies regarding its use in orthopedic trauma surgery. Studies have shown the effectiveness and safety of TXA at FIT, but presented different forms of administration (intravenous, topical, infiltrative) . Despite promising results to contain bleeding in elective orthopedic surgery and fractures, in daily practice, TXA is not very popular, especially in fractures, and has not been used routinely by all doctors. Studies have not been found in the literature about the topical use of TXA compared to intravenous use in FIT.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any sex or skin color older than 60 years, admitted for surgical treatment of FIT with indication of fixation with cephalomedullary nails (PFN) in fractures reduced to closed focus.

Exclusion Criteria:

* hypersensitivity to TXA;

  * Thrombocytopenia and coagulation disorders: platelets <100,000 or prothrombin activity time (TAP) <70% or activated partial thromboplasty time (APTT)> 40 seconds or International Standardized List (INR)> 1;
  * Hepatorenal dysfunction or severe heart disease;
  * Previous surgery in the same place;
  * Use of anticoagulants and corticoids;
  * Pathological fractures of neoplastic origin or duration of neoplastic treatment;
  * Autoimmune disease;
  * History of pulmonary embolism;
  * History of any type of thrombosis (cerebral, in limbs) or stroke;
  * Body Mass Index ≥ 40kg / m2 ;
  * Patients in need of a second surgical access to reduce the fracture with a direct approach to the fracture focus;
  * Diabetes with difficult control.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-12-18 (Estimated); Study Completion 2022-12-18 (Estimated)

PRIMARY OUTCOMES:
To assess bleeding loss in operative intertrochanteric fractures | 2 YEARS
  Blood loss assessment:
  Patients will be evaluated 1 day before surgery and on the first and second postoperative days with the following laboratory tests: complete blood count and coagulogram, hemoglobin, hematocrit, APTT and INR. The calculation of the estimated initial blood volume will be: Women: (height in meters x 0.3561) + (weight in Kg x 0.03308) + 0.1833 and men: (height in meters x 0.3669) + (weight in Kg x 0.03219) + 0.6041(LEVINE et al., 2014; ALMEIDA et al., 2018).
  Blood loss (PS) will be calculated in milliliters (ml), based on the hemoglobin levels adjusted for the patient's initial blood volume. PS = Estimated initial volume x (Initial hematocrit less (-) post-operative hematocrit) / (Initial hematocrit)) (GROSS, 1983).

CONTACTS AND LOCATIONS:
Overall Officials: Carlos DM ARAÚJO, MD, PhD, Principal Investigator — Universidade do Vale do Sapucai
Locations (1):
- Hospital das Clinicas Samuel Libanio, Pouso Alegre, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foss NB, Kehlet H. Hidden blood loss after surgery for hip fracture. J Bone Joint Surg Br. 2006 Aug;88(8):1053-9. doi: 10.1302/0301-620X.88B8.17534. PMID 16877605
- [Background] Henry DA, Carless PA, Moxey AJ, O'Connell D, Stokes BJ, Fergusson DA, Ker K. Anti-fibrinolytic use for minimising perioperative allogeneic blood transfusion. Cochrane Database Syst Rev. 2011 Mar 16;2011(3):CD001886. doi: 10.1002/14651858.CD001886.pub4. PMID 21412876
- [Background] Lei J, Zhang B, Cong Y, Zhuang Y, Wei X, Fu Y, Wei W, Wang P, Wen S, Huang H, Wang H, Han S, Liu S, Zhang K. Tranexamic acid reduces hidden blood loss in the treatment of intertrochanteric fractures with PFNA: a single-center randomized controlled trial. J Orthop Surg Res. 2017 Aug 15;12(1):124. doi: 10.1186/s13018-017-0625-9. PMID 28810918
- [Background] Mohib Y, Rashid RH, Ali M, Zubairi AJ, Umer M. Does tranexamic acid reduce blood transfusion following surgery for inter-trochanteric fracture? A randomized control trial. J Pak Med Assoc. 2015 Nov;65(11 Suppl 3):S17-20. PMID 26878513
- [Background] Tengberg PT, Foss NB, Palm H, Kallemose T, Troelsen A. Tranexamic acid reduces blood loss in patients with extracapsular fractures of the hip: results of a randomised controlled trial. Bone Joint J. 2016 Jun;98-B(6):747-53. doi: 10.1302/0301-620X.98B6.36645. PMID 27235515
- [Background] Zhou XD, Zhang Y, Jiang LF, Zhang JJ, Zhou D, Wu LD, Huang Y, Xu NW. Efficacy and Safety of Tranexamic Acid in Intertrochanteric Fractures: A Single-Blind Randomized Controlled Trial. Orthop Surg. 2019 Aug;11(4):635-642. doi: 10.1111/os.12511. Epub 2019 Aug 16. PMID 31419080
- [Background] Zhu Q, Yu C, Chen X, Xu X, Chen Y, Liu C, Lin P. Efficacy and Safety of Tranexamic Acid for Blood Salvage in Intertrochanteric Fracture Surgery: A Meta-Analysis. Clin Appl Thromb Hemost. 2018 Nov;24(8):1189-1198. doi: 10.1177/1076029618783258. Epub 2018 Jun 21. PMID 29929380
- [Result] Bostrom J, Grant JA, Fjellstrom O, Thelin A, Gustafsson D. Potent fibrinolysis inhibitor discovered by shape and electrostatic complementarity to the drug tranexamic acid. J Med Chem. 2013 Apr 25;56(8):3273-80. doi: 10.1021/jm301818g. Epub 2013 Apr 10. PMID 23521080
- [Result] Diaz AR, Navas PZ. Risk factors for trochanteric and femoral neck fracture. Rev Esp Cir Ortop Traumatol (Engl Ed). 2018 Mar-Apr;62(2):134-141. doi: 10.1016/j.recot.2017.09.002. Epub 2018 Feb 21. English, Spanish. PMID 29429857